CLINICAL TRIAL: NCT01656356
Title: Phase I Safety and Immunogenicity of Live Attenuated Influenza H5 Candidate Vaccine Strain A/17/Turkey/Turkey/05/133 (H5N2) in Healthy Thai Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Punnee Pitisuttithum, Professor, Mahidol University
Other Study IDs: GPO AVIAN FLU Vaccine-V02
Record Dates: First submitted 2012-07-25; First posted 2012-08-03 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Preventive Avian Flu
Keywords: Avian Flu; H5N2
MeSH Terms: conditions — Influenza in Birds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A/17/turkey/Turkey/05/133 (H5N2) (Active Comparator)
  Interventions: Biological: Avian Flu Vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Avian Flu Vaccine
  Arms: A/17/turkey/Turkey/05/133 (H5N2)
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and reactogenicity of live attenuated influenza H5 vaccine candidate strain A/17/turkey/Turkey/05/133 (H5N2) manufactured by GPO, in Thailand to previously healthy Thais.

DETAILED DESCRIPTION:
It is a phase I randomized placebo controlled trial (vaccine and placebo ratio of 2:1). A phase II study is planned to be conducted following review of results of this phase.

Phase I: It is a double blind randomized placebo controlled trial involving 24 participants age 18-49 years (16 will receive vaccines and 8 will receive placebo). All will be admitted in the isolation ward for 10-14 days after each immunization mainly for safety assessment. Two doses of live attenuated influenza H5 vaccine candidate strain A/17/turkey/Turkey/05/133 (H5N2) will be given by intranasal route 21 days apart. Each group of 4 participants will be immunized at a time at 30-60 mins interval. All participants will be followed 21 days after each immunization. Total follow up is 60 day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age 18-49 years old
* Having Thai ID card or equivalent
* Are seronegative to the specific H5 influenza virus determined by antibody titer less than 1:40 by HAI test to the corresponding antigen.
* Anti HIV - Negative
* All hematology & biochemistry and urine analysis are within normal range or of no clinical significance (not more than 1.5 times of normal value)
* Able to read and write and sign written informed consent.

Exclusion Criteria:

* Known history of egg allergy
* Having had recently influenza infection confirmed as H5
* History of bronchial asthma
* History of chronic lung diseases
* History of chronic rhinitis
* History of immunodeficiency state
* History of immunosuppression
* History of heavy smoking (more than 5 rolls per day)
* History of alcoholic (pure drink 200 ml per day)
* Acute infectious and noninfectious diseases (within 2 weeks)
* Exacerbation of chronic diseases or cancer or HIV positives
* Anamnestic leukocytosis, hepatitis B and C positives
* The volunteers who have been taking immunoglobulin products or have had a blood transfusion during past three months before the beginning of the experiment
* Participation in other research study or stop participant less than 1 month
* Pregnancy or plan to become pregnant for 60 days after enrollment or breast feeding
* Any concomitant medication with Aspirin
* The volunteers who have family members with immunodeficiency
* Poultry workers
* Have undertaken international travel within the one week prior to immunization

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2012-05; Primary Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Tropical Medicine, Bangkok, Bangkok, Thailand